CLINICAL TRIAL: NCT01651793
Title: Effect of Phytochemicals From Theobroma Cacao on Mental Energy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: The Hershey Company (Industry)
Responsible Party: Principal Investigator, Patrick O'Connor, Professor of Kinesiology, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Study of cocoa-like beverages
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Mental Fatigue
Keywords: cacao; theobromine; flavanols; caffeine; sustained attention; vigilance; vigor; vitality; energy; fatigue
MeSH Terms: conditions — Mental Fatigue; Fatigue | interventions — Chocolate; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Caffeinated cocoa (Active Comparator): High flavanol, high theobromine, high caffeine, single dose administration in hot water vehicle
  Interventions: Other: Caffeinated cocoa
- Cocoa (Active Comparator): High flavanol, high theobromine, low caffeine, single dose administration in hot water vehicle
  Interventions: Other: Cocoa
- Caffeine (Active Comparator): Low flavanol, low theobromine, high caffeine, single dose administration in hot water vehicle
  Interventions: Other: Caffeine
- Placebo (Placebo Comparator): No flavanol, no theobromine, no caffeine, single dose administration in hot water vehicle
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Caffeinated cocoa — 70 mg caffeine, 179 mg theobromine, 499 mg flavanols, and 1 packet of Truvia sweetener
  Arms: Caffeinated cocoa
Other: Cocoa — 21 mg caffeine, 179 mg theobromine, 499 mg flavanols, and 1 packet of Truvia sweetener
  Arms: Cocoa
Other: Caffeine — 473 ml brewed water containing 66 mg caffeine, caramel coloring and one packet Truvia sweetener
  Arms: Caffeine
Other: Placebo — 473 ml of brewed water, caramel coloring and one packet Truvia sweetener
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine which substances in cocoa produces changes in mental energy. This is a double blind study. The primary outcome measures are performance on tasks of sustained attention (serial subtract, continuous performance test and Bakan task) at pre and 90, 120 and 160 minutes post intervention, energy and fatigue symptoms (profile of mood state), and ratings of motivation to perform cognitive tasks. The assigned interventions are the following:

DETAILED DESCRIPTION:
Only one prior study has examined the acute influence of cocoa on mental energy. The purpose of this research is to replicate the previous observations and extend research in four ways: 1) start to determine which substance in cocoa responsible for the effect by including several comparison groups, 2) focus on individuals with average or below average symptoms of mental energy and who are not high consumers of fruits, vegetables and other products containing high amounts of flavonoids in order to learn whether people with low energy accrue a greater benefit, and 3) include additional measures of mental energy plausibly influenced by cocoa to better understand the health consequences of cocoa.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ages 18-34
* Lower than average feelings of energy (score of < 13 on Profile of Mood States Vigor scale)

Exclusion Criteria:

* Pregnant
* GI tract disorder
* Psychoactive medication use
* Daily consumption of > 200 mg caffeine
* Body mass index > 30
* Cigarette smoker
* Allergy to cocoa, chocolate or caffeine
* Frequent consumption of cocoa, chocolate-based products or fruits and vegetable containing flavonoids

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick O'Connor, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be kept securely at the University of Georgia for several years and can be accessed upon request by contacting Dr. Pat O'Connor (poconnor@uga.edu).
Time Frame: January 1, 2019
Access Criteria: Open Access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited from (i) large university classes, (ii) announcements on buses, bulletin boards, and electronic listservs, and (iii) through word of mouth. Potential participants were invited to complete screening questionnaires (medical history, diet, mood) administered online using Zoomerang
  >http://www.zoomerang.com/<.
Groups:
- Caffeinated Cocoa, Cocoa, Caffeine, Placebo: Order: Caffeinated cocoa, cocoa, caffeine, Placebo; 6 participants were randomized to this order.
- Cocoa, Caffeine, Placebo, Caffeinated Cocoa: Order: Cocoa, Caffeine, Placebo, Caffeinated Cocoa; 6 participants were randomize to receive treatment in this order.
- Caffeine, Placebo, Caffeinated Cocoa, Cocoa: Order: Caffeine, Placebo, Caffeinated cocoa, Cocoa; 6 participants were randomized to receive treatment in this order.
- Placebo, Caffeinated Cocoa, Cocoa, Caffeine: Order: Placebo, Caffeinated cocoa, Cocoa, Caffeine; 6 participants were randomized to receive treatment in this order.
Period: Overall Study
Arm/Group | Caffeinated Cocoa, Cocoa, Caffeine, Placebo | Cocoa, Caffeine, Placebo, Caffeinated Cocoa | Caffeine, Placebo, Caffeinated Cocoa, Cocoa | Placebo, Caffeinated Cocoa, Cocoa, Caffeine
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Completed Participants: These baseline data represent all participants who completed the trial (n = 23). Data are presented as means and standard deviations where appropriate.
Arm/Group | All Completed Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 20 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 15
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23
Amount of sleep on a typical night in the past month (hrs) [Mean (Standard Deviation); unit: hours] | 7.4 (1.1)
Height [Mean (Standard Deviation); unit: cm] | 168.28 (1.19)
Weight [Mean (Standard Deviation); unit: kg] | 67.05 (14.87)

OUTCOME MEASURES:

1. Primary Outcome: Correct Responses on Serial 7 Subtraction Task
Description: Participants subtract the number 7 from a three digit number and quickly and accurately as possible for 60 seconds. The total number of accurate responses is scored. The higher the score the better performance. The range of scores is from a minimum score of 0 to a theoretical maximum score of 120.
Time Frame: Pre and 30, 60 and 120 minutes post intervention
Measure: Mean (Standard Deviation); unit: Correct responses
Groups:
- Pre-test: Baseline measures, pre consumption of beverages.
- Post-test 1: 21-47 minutes post consumption.
- Post-test 2: 57-83 minutes post consumption.
- Post-test 3: 93-119 minutes post consumption.
Arm/Group | Pre-test | Post-test 1 | Post-test 2 | Post-test 3
Number analyzed (Participants) | 23 | 23 | 23 | 23
Correct responses
  Subtract 7 Correct - Placebo | 40.91 (5.56) | 42.57 (3.51) | 43.04 (2.31) | 42.13 (3.67)
  Subtract 7 Correct - Caffeine | 41.83 (3.56) | 41.35 (3.73) | 43.22 (2.92) | 42.74 (3.03)
  Subtract 7 Correct - Cocoa | 42.57 (2.52) | 42.61 (3.86) | 42.78 (3.06) | 42.61 (3.81)
  Subtract 7 Correct - Caffeine + Cocoa | 42.17 (3.24) | 42.26 (2.47) | 42.96 (2.33) | 43.14 (2.88)
Statistical Analysis 1: Comparison: Pre-test; Hypotheses were tested using a series (all outcome variables) of 2 Treatment x 4 Time point, repeated measures ANCOVAs that controlled for the prior night's sleep. Primary interests were the presence of statistically significant interactions of time and either cocoa versus placebo, cocoa + caffeine versus cocoa, or cocoa + caffeine versus caffeine-only. Significant interactions were decomposed using one-way ANOVAs and t-tests with familywise error controlled using LSD post-hoc tests; Test type: Superiority; p = 0.05, ANCOVA — P value reference to the beverage x time interaction effect

2. Primary Outcome: Performance on Bakan Task
Description: Performance on Bakan Task at baseline, post-test 1, post-test 2, and post-test 3
  Bakan test presents numbers on a computer screen. Participant presses one button whenever the number 6 appears and a different button whenever three odd and different numbers in a row occurs such as 7 5 9. The number of times the participant does this correctly the better the performance. The scores range from 0 to 10 because the sequence of three odd and different numbers occurs a total of 10 times.
Time Frame: baseline, post 60, post 90, post 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-test | Post-test 1 | Post-test 2 | Post-test 3
Number analyzed (Participants) | 23 | 23 | 23 | 23
units on a scale
  Bakan Primary Correct - Placebo | 6.35 (1.53) | 6.00 (1.57) | 5.96 (2.01) | 6.09 (1.95)
  Bakan Primary Correct - Caffeine | 6.35 (1.50) | 6.57 (1.78) | 6.87 (1.39) | 6.13 (1.36)
  Bakan Primary Correct - Cocoa | 6.43 (1.59) | 6.52 (1.44) | 6.30 (1.11) | 5.78 (1.70)
  Bakan Primary Correct - Caffeine + Cocoa | 5.83 (1.59) | 6.13 (1.77) | 6.35 (1.77) | 6.61 (1.47)

3. Secondary Outcome: Vigor Symptoms (Profile of Mood State)
Description: Vigor subscale scores from the Profile of Mood States.The higher the score the greater the feelings of energy. The scores range from a minimum of 0 to a maximum of 20.
Time Frame: Pre and 90, 120 and 160 minutes post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pre-test: Mood measure at baseline.
- Post-test 1: 22-48 minutes post consumption.
- Post-test 2: 60-86 minutes post consumption.
- Post-test 3: 98-124 minutes post consumption.
Arm/Group | Pre-test | Post-test 1 | Post-test 2 | Post-test 3
Number analyzed (Participants) | 23 | 23 | 23 | 23
units on a scale
  POMS Vigor - Placebo | 3.78 (4.36) | 3.57 (4.00) | 3.52 (3.44) | 3.65 (3.68)
  POMS Vigor - Caffeine | 3.91 (3.66) | 3.91 (3.99) | 4.00 (3.92) | 4.26 (3.29)
  POMS Vigor - Cocoa | 3.65 (4.01) | 3.74 (3.45) | 4.00 (3.84) | 3.70 (3.30)
  POMS Vigor - Caffeinated Cocoa | 4.09 (4.43) | 4.48 (4.28) | 4.04 (4.03) | 4.17 (3.87)

ADVERSE EVENTS:
Time Frame: The study personnel monitored participants through study completion, an average of 4 weeks, for adverse events. No adverse events were reported to study personnel.
Groups:
- Caffeinated Cocoa: High flavanol, high theobromine, high caffeine, single dose administration in hot water vehicle
  Active comparator 1: High flavanol, high theobromine, high caffeine, single dose administration in hot water vehicle
- Cocoa: High flavanol, high theobromine, low caffeine, single dose administration in hot water vehicle
  Active comparator 2: High flavanol, high theobromine, low caffeine, single dose administration in hot water vehicle
- Cafeine: Low flavanol, low theobromine, high caffeine, single dose administration in hot water vehicle
  Active comparator 4: Low flavanol, low theobromine, high caffeine, single dose administration in hot water vehicle
- Placebo: No flavanol, no theobromine, no caffeine, single dose administration in hot water vehicle
  Inactive comparator: No flavanol, no theobromine, no caffeine, single dose administration in hot water vehicle
Arm/Group | Caffeinated Cocoa | Cocoa | Cafeine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
Recruitment targeted those reporting low consumption of fruits and vegetables and other foods containing flavonols; not all participants were medication-free; the potential role of sensory aspects of cocoa were not examined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes